CLINICAL TRIAL: NCT01430247
Title: Vision Screening of the Four Year Old Children for the Detection of Amblyopia in The Town of Zagreb
Brief Title: Vision Screening for the Detection of Amblyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mladen Busic (Other)
Responsible Party: Sponsor-Investigator, Mladen Busic, Asst. prof., M.D., PhD, General Hospital Sveti Duh
Organization: General Hospital Sveti Duh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 30082011/2011
Record Dates: First submitted 2011-08-31; First posted 2011-09-08 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Amblyopia; Refractive Errors; Anisometropia; Strabismus; Ptosis
Keywords: amblyopia; amblyogenic factors; screening; preschool children; visual acuity; prevalence
MeSH Terms: conditions — Amblyopia; Refractive Errors; Anisometropia; Strabismus; Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amblyopia screening (Other)
  Interventions: Other: Amblyopia screening

INTERVENTIONS:
Other: Amblyopia screening — Monocular vision testing at near (40cm) and distance (3m)

SUMMARY:
INTRODUCTION. Amblyopia is defined as the loss of visual acuity (VA) in one or both eyes, without any obvious structural or pathological anomalies. Amblyopic eye should be able to regain some VA if treatment is initiated before the age of seven. It is the leading cause of monocular blindness in the 20- to 70-year olds with prevalence 2-5%. Amblyopia is mainly monocular, hence children are general asymptomatic. VA testing is the only reliable method of detecting amblyopia, and the fourth year of life is considered best for vision screening programs.

AIM: The purpose of the study is to reduce the preventable vision loss. The main goal of the study is to evidence the problem of amblyopia in Zagreb and to release a model for formal, government directed vision-screening program as a Croatian public health policy.

HYPOTHESIS. In Croatia, the prevalence and actual effect of amblyopia and amblyogenic factors, along with treatment efficacy is impossible to quantify, since no population-based studies have been performed regarding this issue. In addition, national screening of preschool children does not exist, while the school-entry screening is prescribed by law. The object of the study is to determine the prevalence of amblyopia in a 4-4.5 year old children of The Town of Zagreb, the efficacy of screening and effectiveness of treatment on reducing amblyopia prevalence. The primary hypothesis is defined: screening of visual acuity monocularly at distance and near in 4-4.5 year old children in Zagreb is effective in detecting amblyopia.

PATIENTS AND METHODS: Monocular vision of about 7000 children/ year aged 4-4.5 for whom both parents gave consent is to be tested with Lea chart at near (40cm) and distance (3m) in the kindergartens of The Town of Zagreb. The criterion for referral to complete ophthalmological examination is VA <0.8.

ELIGIBILITY:
Inclusion Criteria:

* children in the kindergartens of The Town of Zagreb aged 4-4.5 for whom both parents gave written informed consent

Exclusion Criteria:

* children younger than 4 years and children older than 4.5 years

Ages: 48 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7000 (Actual)
Dates: Start 2011-09-12 (Actual); Primary Completion 2014-09-12 (Actual); Study Completion 2014-09-12 (Actual)

PRIMARY OUTCOMES:
prevalence of amblyopia | 3 years
  proportion of children with amblyopia in a total population of children screened

CONTACTS AND LOCATIONS:
Overall Officials: Mladen Bušić, Principal Investigator — University Eye Clinic, University Hospital "Sveti Duh", Zagreb, Croatia
Locations (1):
- University Eye Clinic, University Hospital "Sveti Duh", Zagreb, Croatia